CLINICAL TRIAL: NCT04460300
Title: The Effect of Aromatherapy Through Inhalation and Foot Massage on Blood Pressure and Stress Response in Individuals With Essential Hypertension
Brief Title: Effects of Aromatherapy in Hypertensive Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AIBU-HSF-SCC-02
Record Dates: First submitted 2020-06-21; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Essential Hypertension; Aromatherapy; Stress, Physiological
Keywords: Essential Hypertension; Aromatherapy; Physiological Stress Response; Anxiety; Arterial Pressure
MeSH Terms: conditions — Essential Hypertension; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aromatherapy-inhalation group (Experimental): In addition to the pharmacological treatment prescribed by the physician to individuals in this group, aromatherapy is carried out through the essential oil inhalation method. Individuals who can distinguish odors in the odor sense test before the application is included in the study. Aromatherapy inhalation is applied for three days and every other day (eg Monday-Wednesday-Friday) determined by the researchers for a week. Intervention is made between 07:00 and 08:00 in the morning hours when the blood cortisol value is maximized and homogeneity is provided.
  In this method, 5 drops of lavender oil is dropped directly on a sterile gauze and individuals is allowed to breathe from a distance of 10 cm for 5 minutes.
  Interventions: Other: Aromatherapy-inhalation method
- Aromatherapy-foot massage group (Experimental): In addition to the pharmacological treatment prescribed by the physician to individuals in this group, aromatherapy is applied through foot massage. Swedish massage protocol is followed in foot massage intervention.The foot massage is performed on three days and every other day (eg Monday-Wednesday-Friday) determined by the researchers for a week.The intervention is performed between 07:00 and 08:00 in the morning hours when the blood cortisol value is maximized and homogeneity is provided.
  Foot massage is done with 10 drops (5 drops per foot) of lavender for 10 minutes for each foot for 20 minutes. During the intervention, 20 techniques is used and the application time of each technique is 30 seconds (total 10 minutes per foot).
  Interventions: Other: Aromatherapy-foot massage group
- Control group (No Intervention): Interviews is held with the control group while performing the routine treatment and care of the clinic. No intervention is made by the researchers to the control group during the interview.

INTERVENTIONS:
Other: Aromatherapy-inhalation method — In addition to the pharmacological treatment prescribed by the physician to individuals in this group, aromatherapy is carried out through the essential oil inhalation method. Individuals who can distinguish odors in the odor sense test before the application is included in the study. Aromatherapy inhalation is applied for three days and every other day (eg Monday-Wednesday-Friday) determined by the researchers for a week. Intervention is made between 07:00 and 08:00 in the morning hours when the blood cortisol value is maximized and homogeneity is provided.
  In this method, 5 drops of lavender oil will be dropped directly on a sterile gauze and individuals will be allowed to breathe from a distance of 10 cm for 5 minutes.
  Arms: Aromatherapy-inhalation group
Other: Aromatherapy-foot massage group — In addition to the pharmacological treatment prescribed by the physician to individuals in this group, aromatherapy is applied through foot massage. Swedish massage protocol is followed in foot massage intervention.The foot massage is performed on three days and every other day (eg Monday-Wednesday-Friday) determined by the researchers for a week.The intervention is performed between 07:00 and 08:00 in the morning hours when the blood cortisol value is maximized and homogeneity is provided.
  Foot massage is done with 10 drops (5 drops per foot) of lavender for 10 minutes for each foot for 20 minutes. During the intervention, 20 techniques is used and the application time of each technique is 30 seconds (total 10 minutes per foot).
  Arms: Aromatherapy-foot massage group

SUMMARY:
Objective: To investigate the effect of aromatherapy on blood pressure and stress response by inhalation and foot massage in individuals with essential hypertension.

Methods: The randomized controlled trial is performed with 69 individuals diagnosed with essential hypertension hospitalized. There are two interventions (group 1: aromatherapy-inhalation method, group 2: aromatherapy-foot massage) and a control group in the study. Blood pressure is measured with a digital sphygmomanometer after 10 minutes of rest; stress response is determined by heart rate, blood cortisol levels and anxiety scale. Aromatherapy with lavender oil is applied to the intervention groups; no application is made to the control group and routine follow-up at the hospital continued.

DETAILED DESCRIPTION:
Objective: The primary aim of the study is to investigate the effect of aromatherapy on blood pressure and stress response by inhalation and foot massage in individuals with essential hypertension. Secondary aims;

* to define the effect of aromatherapy inhalation method and foot massage application on blood pressure and heart rate in individuals with essential hypertension,
* to define the effects of aromatherapy inhalation method and foot massage application on blood cortisol levels in individuals with essential hypertension,
* to define the effects of aromatherapy inhalation method and foot massage application on anxiety scores in individuals with essential hypertension.

Hypothesis:

* H0-1: Aromatherapy inhalation method has no significant effect on blood pressure in individuals with essential hypertension.
* H1-1: Aromatherapy inhalation method has a significant effect on blood pressure in individuals with essential hypertension.
* H0-2: Aromatherapy inhalation method does not have a significant effect on stress response in individuals with essential hypertension.
* H1-2: Aromatherapy inhalation method has a significant effect on stress response in individuals with essential hypertension.
* H0-3: Foot massage application does not have a significant effect on blood pressure in individuals with essential hypertension.
* H1-3: Foot massage application has a significant effect on blood pressure in individuals with essential hypertension.
* H0-4: Foot massage application in patients with essential hypertension has no significant effect on stress response.
* H1-4: Foot massage application in patients with essential hypertension has a significant effect on stress response.

Methods: The randomized controlled trial is performed with 69 individuals diagnosed with essential hypertension hospitalized.There are two interventions (group 1: aromatherapy-inhalation method, group 2: aromatherapy-foot massage) and a control group in the study. In power analysis based on blood cortisol level,80% power, 95% confidence interval, effect size 0.39, standard deviation 3.09 were calculated and 23 participants in each group were determined. Blood pressure is measured with a digital sphygmomanometer after 10 minutes of rest; stress response is determined by heart rate, blood cortisol levels and anxiety scale. Aromatherapy with lavender oil is applied to the intervention groups; no application is made to the control group and routine follow-up at the hospital continued. The group-1 smells sterile cloth with 5 drops of lavender oil for five minutes and is done every other day for three days. Group-2 receives a total of 20 minutes of foot massage with 5 drops of lavender oil for each foot and is applied every other day for three days. Aromatherapy is performed between 07:00 and 08:00 in the morning hours when the blood cortisol value peaked at the highest level and homogeneity is achieved in terms of application.

Measures: For intervention groups (group 1 and 2), blood pressure and heart rate will be measured seven times in total, both at the first interview and before and after each application, 10 minutes after the application; for control group, it is a total of seven times, both once in the first interview and twice every other day. Blood cortisol level is measured four times in total for the intervention groups, both at the beginning and after each application; For the control group, it is measured at the same time as the intervention groups at baseline and on the third follow-up day (twice in total). Anxiety scale (Spielberger State-Trait Anxiety Inventory) is used for subjective stress response. Trait Anxiety Inventory is evaluated at the beginning of the study for both groups (only once). State Anxiety Inventory, for intervention groups, is applied four times both before and after the first application and before and after the third application; for control group is applied twice, on the first follow-up day and on the third follow-up day.

Analysis: Statistical methods to be used for study data;

* Descriptive statistics (number and percentage, average, standard deviation)
* T test (Parametric), Mann Whitney U test (nonparametric) (according to the suitability of the data for normal distribution)
* One-way anova (Parametric), Kruskal Wallis Test (nonparametric) (according to the normal distribution of data)
* Pearson / Spearman Correlation (according to the suitability of the data for normal distribution)
* Analysis of variance in repeated measurements
* Regression analysis

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* Have been diagnosed with essential hypertension for at least 6 months,
* Blood pressure values are 120-180 mmHg for systolic pressure and 80-110 mmHg for diastolic pressure,
* Receiving regular antihypertensive therapy,
* No additional antihypertensive drug is added during the application,
* Passing the odor sense test,
* No current anxiolytic or hypnotic treatment,
* Not diagnosed with psychiatric illness,
* Not pre-applied,
* Those who understand and speak Turkish,
* No speech, hearing and vision loss,
* Non-smoker,
* Does not apply herbal treatment to lower blood pressure,
* Individuals who agreed to participate in the research

Exclusion Criteria:

* An additional antihypertensive drug was added during the application,
* Before each intervention, SKB ≥ 180 or <120 mmHg and DKB ≥ 110 or <80 mmHg,
* Taking dialysis treatment,
* In addition to its existing diseases, it is diagnosed with asthma, COPD and acute myocardial infarction.
* With a known allergic response to lavender oil,
* Applying herbal treatment to lower blood pressure,
* Those who cannot pass the odor sense test,
* Receiving current anxiolytic or hypnotic treatment,
* Diagnosed with psychiatric illness,
* Pre-implemented,
* Who cannot understand and speak Turkish,
* Speech, hearing and vision loss,
* Smoker,
* Individuals who do not agree to participate in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2018-12-03 (Actual); Primary Completion 2020-08-03 (Estimated); Study Completion 2020-08-03 (Estimated)

PRIMARY OUTCOMES:
Mean of blood pressure (mmHg) | up to one week
  In the study, a digital sphygmomanometer, which has been calibrated in comparison with the mercury sphygmomanometer, is used in order to prevent individual differences in the measurement of blood pressure. For accurate results, the sphygmomanometer sleeve is sized for adult individuals (width = about 20 cm, length = about 40 cm). In order for the blood pressure not to be affected by the conditions during the measurement, it is taken into account that the individual did not drink tea or coffee, take caffeine, and preferably did not eat during the 30 minutes prior to measurement. Measurements are made after the individual has been resting in a quiet room for at least 10 minutes. The measurements at the first interview are made from both arms, the blood pressure in the high arm is considered to be the blood pressure of the patient. Blood pressure measurements in the follow-ups are also made from this arm.
Mean of heart rate (/dk) | up to one week
  The heart rate is the pressure of the left ventricle on the vascular wall of the blood that it throws into the aorta during systole from the skin surface.In the research, apical heart rate is measured with a stethoscope.
Mean of blood cortisol level (mg/dl) | up to one week
  Adrenal cortisol release is largely regulated by the limbic system-hypothalamus-pituitary and adrenal (L-HPA) axis.When an individual detects an environmental stimulus or stress to be avoided, activation of the HPA-axis is initiated in the central nervous system, and a physiological process occurs to stimulate the adrenal gland to release glucocorticoids for cortisol release.There are sources showing that the maximum cortisol values are between 04:00 and 08:00. The half-life of cortisol in circulation is 60 minutes, so the blood concentration changes rapidly. For this reason, interventions in the study are performed within hours when the serum cortisol level is highest and blood will be drawn for cortisol 5 minutes after the application.
Means of subjective anxiety scores | up to one week
  Spielberger State-Trait Anxiety Inventory is used to measure subjective anxiety scores.The State Anxiety Inventory is a 4-point Likert-type scale consisting of 20 questions aimed at measuring how individuals are feeling right now.The Trait Anxiety Inventory is a 20-item scale that generally determines how the individual feels, regardless of the situation and circumstances in which the individual is present.

CONTACTS AND LOCATIONS:
Overall Officials: Saadet Can Cicek, Principal Investigator — Bolu Abant Izzet Baysal University, Health Sciences Faculty
Locations (1):
- Bolu Elderly Health Center, Bolu, Turkey (Türkiye)

REFERENCES:
- [Derived] Can Cicek S, Demir S, Yilmaz D, Acikgoz A, Yildiz S, Yis OM. The Effect of Aromatherapy on Blood Pressure and Stress Responses by Inhalation and Foot Massage in Patients With Essential Hypertension: Randomized Clinical Trial. Holist Nurs Pract. 2022 Jul-Aug 01;36(4):209-222. doi: 10.1097/HNP.0000000000000526. PMID 35708557